CLINICAL TRIAL: NCT02865590
Title: Clinical and Histological Evaluation of Demineralized Bone Allograft and Lyophilized Equine Bone Allograft for Sinus Lift: Double Blind, Parallel, Randomized Clinical Trial.
Brief Title: Clinical and Histological Evaluation of Deproteinizated Bovine Bone Allograft and Lyophilized Equine Bone Allograft for Sinus Lift.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Enrico Marchetti, assistant professor, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Prot.001/luglio2010
Record Dates: First submitted 2015-10-03; First posted 2016-08-12 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Maxillary Sinus Floor Augmentation
Keywords: Maxillary Sinus/surgery; Bone Substitutes; Radiography, Panoramic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lyophilized Equine Bone Allograft (Experimental): Sinus Lift with Lyophilized Equine Bone Allograft
  Interventions: Device: sinus lift with Lyophilized Equine Bone Allograft (Bio-gen , Bioteck s.p.a., Arcugnano (VI) - Italy)
- deproteinized bovine bone allograft (Active Comparator): Sinus lift with deproteinized bovine bone allograft
  Interventions: Device: Sinus lift with deproteinized bovine bone allograft (Endobon Xenograft Granules, Zimmer Biomet, San Donato Milanese (MI) - Italy)

INTERVENTIONS:
Device: sinus lift with Lyophilized Equine Bone Allograft (Bio-gen , Bioteck s.p.a., Arcugnano (VI) - Italy)
  Arms: Lyophilized Equine Bone Allograft
Device: Sinus lift with deproteinized bovine bone allograft (Endobon Xenograft Granules, Zimmer Biomet, San Donato Milanese (MI) - Italy)
  Arms: deproteinized bovine bone allograft

SUMMARY:
The sinus infiltration technique for sinus floor elevation has been used successfully when a reduced vertical height is available in the posterior maxilla. However, the effect of the different graft material on the volume and on the quality of new bone formed has not been fully investigated. The aim of this study is to evaluate the clinical and histological effect of a test material, lyophilized equine bone (Bio-gen®), compared with control material, deproteinized bovine bone (Endobon®), in the sinus lift techniques with lateral approach.

ELIGIBILITY:
Inclusion Criteria:

* bilateral atrophy of the maxilla;
* bone ridge <= 6mm

Exclusion Criteria:

* severe systemic diseas (ASA III -IV) bisphosphonate therapy or a history of up to 3 years history of radiation therapy to neck and head area sinusitis pregnancy subjects not able to consent to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GIUSEPPE MARZO, DMD, Study Chair — University of L'Aquila

RESULTS

PARTICIPANT FLOW:
Groups:
- Lyophilized Equine Bone Allograft: Sinus Lift with Lyophilized Equine Bone Allograft
  sinus lift with Lyophilized Equine Bone Allograft (Bio-gen , Bioteck s.p.a., Arcugnano (VI) - Italy)
- Deproteinized Bovine Bone Allograft: Sinus lift with deproteinized bovine bone allograft
  Sinus lift with deproteinized bovine bone allograft (Endobon Xenograft Granules, Zimmer Biomet, San Donato Milanese (MI) - Italy)
Period: Overall Study
Arm/Group | Lyophilized Equine Bone Allograft | Deproteinized Bovine Bone Allograft
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 16 patients with a residual crest height of 4 mm or less.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lyophilized Equine Bone Allograft | Deproteinized Bovine Bone Allograft | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Caucasian patients with a residual crest height ≤4 mm who need sinus lift augmentation for dental implant placement.
  Enrolled patients were randomly assigned either to DEBM or AAB groups by a software (STATA/12.1, StataCorp LLC, College Station, TX, USA).
  years | 51 (6.00) | 51 (6.00) | 51 (6.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  Italy | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Histomorphometric Evaluation of New Bone Formation.
Time Frame: 6 months
Population: Caucasion patients aged ≥ 25 years with at least one atrophic posterior maxilla (distally from first bicuspid teeth) with a residual crest height ≤4 mm who need sinus lift augmentation for dental implant placement were eligible for the study.
Measure: Mean (Standard Deviation); unit: percentage of millimeters
Arm/Group | Lyophilized Equine Bone Allograft | Deproteinized Bovine Bone Allograft
Number analyzed (Participants) | 8 | 8
percentage of millimeters
  newly formed bone | 22.20 (7.18) | 22.84 (7.34)
  marrow spaces | 50.77 (7.59) | 46.20 (14.30)
  residual graft material | 27 (6.75) | 30.94 (10.20)

ADVERSE EVENTS:
Arm/Group | Lyophilized Equine Bone Allograft | Deproteinized Bovine Bone Allograft
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No